CLINICAL TRIAL: NCT01820494
Title: Nutritional Management of Infants With Chronic Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AJ85
Record Dates: First submitted 2013-03-26; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Growth and Tolerance Infant Study
Keywords: growth; infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Infant Formula (Experimental): Complete amino acid-based infant formula
  Interventions: Other: Experimental Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — Infant formula to be fed ad libitum
  Other Names: EleCare

SUMMARY:
The study objective is to assess the growth of infants fed an experimental formula for the nutritional management of chronic diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 12 months of age at enrollment
* Candidates for elemental feeding
* Chronic diarrhea and diagnosis of one of the following conditions: short-bowel syndrome, eosinophilic gastroenteritis, food allergy, inflammatory bowel disease, pancreatic disease, protein maldigestion, HIV-advanced disease or other GI disease requiring an elemental diet or have underlying GI disease without chronic diarrhea if his/her chronic diarrhea is controlled or is in remission by a semi-elemental or elemental formula for no more than 13 weeks
* Parents agree to feed infant with experimental formula for least 50% of total calories during study period

Exclusion Criteria:

* Any non-approved concomitant study

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2000-10; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Weight | Study Day (SD) 1, 28 and 84
  Change in weight from baseline.

SECONDARY OUTCOMES:
Stool Characteristics | Study Day (SD) 2-4, 5-7, 25-27 and 81-83
  Parent completed diary of stool consistency, frequency/volume.

OTHER OUTCOMES:
Dietary Assessment | Study day (SD) 2-4, 5-7, 25-27 and 81-83
  Parent completed record of infant dietary intake.
Blood Chemistry | Study Day (SD) 1 and 84
  Hemoglobin, hematocrit, serum albumin, total protein, urea nitrogen, alkaline phosphatase
Physician Assessment of Abdominal Complaints | Study Day (SD) 1, 28 and 84
  Individualized per subject, may include decreased vomiting, stool number or volume or increased weight gain.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, PhD, RD, Study Chair — Abbott Nutrition
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital of Detroit, Detroit, Michigan
  - Children's Hospital, Omaha, Nebraska

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765
- [Derived] Borschel MW, Antonson DL, Murray ND, Oliva-Hemker M, Mattis LE, Kerzner B, Tolia V, Baggs G. Two single group, prospective, baseline-controlled feeding studies in infants and children with chronic diarrhea fed a hypoallergenic free amino acid-based formula. BMC Pediatr. 2014 May 29;14:136. doi: 10.1186/1471-2431-14-136. PMID 24885833